CLINICAL TRIAL: NCT05270200
Title: To Evaluate Safety and Efficiency of AZA Combined With Chidamide as Maintenance Therapy in High-risk Acute Myeloid Leukemia Patients After Allogeneic Hematopoietic Stem Cell Transplantation：A Multicenter, Single-arm Study
Brief Title: Single Arm Study of Post-transplant Azacitidine and Chidamide for Prevention of Acute Myelogenous Leukemia Relapse
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA+Chidamide
Record Dates: First submitted 2022-01-20; First posted 2022-03-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute myelogenous leukemia; Allogenetic stem cell transplant; Maintenance therapy; Azacitidine; Chidamide; High-risk AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine combined with Chidamide (Experimental): Patients will recieve six courses of azacitidine 50mg/m2 through a needle under your skin on Days 1-3.Each course is 28 days long.At the same time patients will recieve oral chidamide 5mg per day for no more than 2 years.
  Interventions: Drug: Azacitidine; Drug: Chidamide

INTERVENTIONS:
Drug: Azacitidine — Patients will recieve six courses of azacitidine 50mg/m2 through a needle under skin on Days 1-3.Each course is 28 days long.
  Other Names: 5-Azacitidine; 5-aza; Vidaza; 5-AZC
Drug: Chidamide — Patients will recieve oral chidamide 5mg per day for no more than 2 years.
  Other Names: Epidaza

SUMMARY:
The goal of this clinical research study is to learn if azacitidine combined with Chidamide will help to control the disease in patients with high-risk AML after an allogeneic stem cell transplant. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Azacitidine is designed to block certain genes in cancer cells whose job is to stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

Chidamide exhibits potent inhibitory effect on cell viability of MDS and AML cells, and the possible mechanism may lie in the downregulation of JAK2/STAT3 signaling through SOCS3 upregulation.

Study Group： If you are found to be eligible to take part in this study,you will receive azacitidine and chidamide.

Study Drug Administration:

You will recieve six courses of azacitidine through a needle under your skin on Days 1-3.Each course is 28 days long.At the same time you will recieve oral chidamide per day for no more than 2 years.

The treatment will start after 30 days post-transplantation and your neutrophil count is of 1.5 × 10⁹ cells per L or higher and non-transfused platelets is of 80 × 10⁹ per L or higher.

The treatment would stop if neutrophil count is less than 0.5 × 10⁹ cells per L or platelets is less than 50 × 10⁹ per L.And it would also stop when grade 3/4 non-hematological adverse events happened.

Study Visit:

You may come back for study visits every month in a year when the treatment start.

Blood and urine will be drawn for routine tests every month. At 1,2,3,4,5,6,9 and 12 months,You will have a bone marrow aspiration to check the status of the disease.

You will have a electrocardiiogram test every 3 months to check the heart function.

Length of Study:

You will be on study treatment for up to 1 year.You will be taken off study early if you experience intolerable side effects or the disease gets worse.

End-of-Treatment Visit:

If you complete the planned treatment with azacitidine and chidamide, you will have an end-of-treatment visit:

Blood and urine will be drawn for routine tests. You will have a bone marrow aspiration to check the status of the disease. You will have a electrocardiiogram test every 3 months to check the heart function.

This is an investigational study. Azacitidine and chidamide are FDA approved and are commercially available for the treatment of acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age 18 to 60 years old,both male and female
* 2.Be able to understand and sign informed consent
* 3.Patients with a diagnosis of AML not M3 according to the 2016 World Health Organization (WHO) Acute Myeloid Leukemia Classification and Diagnostic
* 4.Patients have AML with poor genetic abnormalities,primary refractory AML,relapsed AML or secondary AML
* 5.Patients with an ECOG performance status 0,1,2 or 3
* 6.Expected survival time ≥ 3 months
* 7.Non-hematological toxicity related to transplantation does not exceed Grade 2
* 8.Laboratory indicators meet the following standards:

  1. 7 days before the first day of the first course of treatment, bilirubin, ALT and AST were all less than 3 times the upper limit of normal.
  2. Measure twice within 7 days before the first day of the first course of treatment, at least 2 days apart, the neutrophil count are greater than 1.5×10/L and without G-CSF treatment.
  3. Measure twice within 7 days before the first day of the first course of treatment, at least 2 days apart, platelet count greater than 80×10/L and without platelet transfusion.
  4. Serum creatinine clearance rate is greater than 30ml/min.

Exclusion Criteria:

* 1.Uncontrollable active infection
* 2.Patients with active hepatitis B or C or HIV infection before enrollment
* 3.Have a grade III-IV graft-versus-host disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Paticipants With Adverse Events as a Measure of Safety | From the day of stem cell transplantation to one year after stem cell transplantation
  Safety were measured with respect to:
  1. Safety measurements
  2. Incidence of adverse events
One year cumulative incidence of relapse | From the day of stem cell transplantation to one year after stem cell transplantation
  Leukemia relapse base on morphoogy criterion

SECONDARY OUTCOMES:
Relapes-free Survival（RFS） | From the day of stem cell transplantation to one year after stem cell transplantation
  The time that a participant survives without relapes of the disease
Overall survival（OS） | From the day of stem cell transplantation to one year after stem cell transplantation
  The time that a participant survives without death
The cumulative Incidence rate of GVHD | From the day of stem cell transplantation to one year after stem cell transplantation
  acute GVHD and chronic GVHD diagnosis based on MIH criterion

OTHER OUTCOMES:
Single-cell sequencing | Before the maintenance therapy and before the 7 cycles of maintenance
  Single-cell sequencing was used to explore the potential mechanism of AZA combined with sidarbenamide to prevent recurrence after transplantation in patients with AML

CONTACTS AND LOCATIONS:
Overall Officials: Rui Huang, Doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Nanfang Hospital of Southern Medical University, Guanzhou, Guandong, China

IPD SHARING:
Plan to Share IPD: Yes
We will share our data within 6 months after the end of the trial. You can ask us for data or obtain it on the Clinical Trial Management Public Platform of clinical trial.
Supporting Information: Study Protocol
Time Frame: The data will be available and permanently disclosed within 6 months after the trial.
Access Criteria: You can log in to the website for data access or contact us for data.